CLINICAL TRIAL: NCT04389697
Title: Fasting Versus Non-Fasting for Cardiac Implantable Electronic Devices (FastCIED Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Health Institute GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019-0310
Record Dates: First submitted 2019-12-20; First posted 2020-05-15 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Cardiac Implantable Electronic Devices

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Clear fluids and food up to up to 1 hour before the procedure
  Interventions: Dietary Supplement: Clear fluids and food up to up to 1 hour before the procedure
- Control arm (No Intervention): Fasting for solids for up to 6 hours and fluids up to 2 hours before the procedure

INTERVENTIONS:
Dietary Supplement: Clear fluids and food up to up to 1 hour before the procedure — Clear fluids and food up to up to 1 hour before the start of the procedure
  Arms: Intervention arm

SUMMARY:
There was no evidence to suggest that a shortened fluid fast results in an increased risk of aspiration, regurgitation or related morbidity compared with the standard 'nil by mouth from midnight' fasting policy. However, there is no available data regarding the safety and efficacy of fasting approach in patients undergoing cardiac implantable electronic device (CIED) procedures. The aim of this study is to demonstrate that a non-fasting protocol is non-inferior in regard to safety to a fasting protocol (current practice) in patients undergoing cardiac device implantation procedures

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years undergoing elective implantation or generator exchange of cardiac implantable electronic devices

Exclusion Criteria:

* Patients presenting with an acute unstable condition (bradycardia < 30/min or temporary pacing wire)
* Patients scheduled for deep sedation
* Patients with increased intra-abdominal pressure (severe intra-abdominal tumors, severe ascites, very severe obesity: BMI>40 kg/m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-12-06 (Actual)

PRIMARY OUTCOMES:
Patients well-being | During the first 24 hours after the procedure
  Post-interventional patients well-being including (to be assessed by questionnaire with the help of a Numeric Rating Scale (rang: 0-10, higher scores mean a worse outcome): abdominal pain, thirst, mouth dryness, headache, anxiety, hunger, nausea, vomiting, tiredness and weakness, dizziness Incidence of Intra -procedural adverse events like emergency intubation and perioperative pulmonary aspiration vomiting)

SECONDARY OUTCOMES:
Usages of inotropic and vasopressor agents | During the intervention
  Amount of used inotropic and vasopressor agents during the intervention
Usage of sedatives | During the intervention
  Amount of used sedative agents during the intervention
Usage of analgesics | During the intervention
  Amount of used analgesics agents during the intervention
Usage anti-vomiting agents | During the intervention
  Amount of used anti-vomiting agents during the intervention
Serum creatinine level | 1 hour pre-procedural, during the first 24 hours after the procedure
  Serum creatinine (mg/dL)
Serum urea level | 1 hour pre-procedural, during the first 24 hours after the procedure
  Serum urea (mg/dL)
eGFR | 1 hour pre-procedural, during the first 24 hours after the procedure
  GFR is Glomerular Filtration Rate and it is a key indicator of renal function. eGFR is estimated GFR and is a mathematically derived entity based on a patient's serum creatinine level, age, sex and race.
Heart rate | pre-intervention, and then every 15 minutes during the procedure
  Heart rate (frequency per minute) will be assessed by using a monitoring device
Oxygen saturation | pre-intervention, and then every 15 minutes during the procedure
  Oxygen saturation (%) will be assessed by using a monitoring device
Blood pressure | pre-intervention, and then every 15 minutes during the procedure
  Systolic and diastolic blood pressure (mmHg) will be assessed by using a monitoring device
blood pH | 1 hour pre-procedural
  Will be assessed by venous blood gas analysis (number).
blood PaCo2 | 1 hour pre-procedural
  Will be assessed by venous blood gas analysis (mmHg).
blood HCO3 | 1 hour pre-procedural
  Will be assessed by venous blood gas analysis (mEq/L).
blood sugar | 1 hour pre-procedural, pre-intervention, 8 hours after procedure
  Will be assessed by venous blood gas analysis (mg/dL).
Sodium | 1 hour pre-procedural, pre-intervention, 8 hours after procedure
  Will be assessed by blood test.
Potassium | 1 hour pre-procedural, pre-intervention, 8 hours after procedure
  Will be assessed by blood test (mm/L).
Patients general satisfaction | During the first 24 hours after the procedure
  Patients general satisfaction with procedure as assessed by the patient satisfaction survey form using Numeric Rating Scale (rang: 0-10, higher scores mean a better outcome)
Sleep quality | During the first 24 hours after the procedure
  Sleep quality based on Numeric Rating Scale (rang: 0-10, higher scores mean a better outcome)
Surgical site pain | During the first 24 hours after the procedure
  Surgical site pain based on Numeric Rating Scale (rang: 0-10, higher scores mean a worse outcome)
Length of ICU stay | Up to 30 days
  Based on the number of ICU stay nights
Length of hospital stay | Up to 30 days
  Based on the number of ICU stay nights plus ward stay
Operation site infection rate | During 30 days after the procedure
  Operation site (Chest) infection rate via Telephone /follow-up visits
Incidence of death | During 30 days after the procedure
  The investigators will then divide the causes into 1) operation related and 2) non-operation related causes

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Bode, MD, MSc, Principal Investigator — Heart Center Leipzig at the University of Leipzig; Alireza Sepehri Shamloo, MD, Principal Investigator — Heart Center Leipzig at the University of Leipzig; Gerhard Hindricks, MD, Study Chair — Heart Center Leipzig at the University of Leipzig
Locations (1):
- Department of Electrophysiology, Leipzig Heart Center, Leipzig, Saxony, Germany

REFERENCES:
- [Derived] Bode K, Gerhards M, Doering M, Lucas J, Tijssen J, Dagres N, Hilbert S, Richter S, Nedios S, Lurz J, Moscoso-Luduena C, Arya A, Shamloo AS, Hindricks G. A randomized trial of non-fasting vs. fasting for cardiac implantable electronic device procedures (Fast-CIED Study). Europace. 2022 Oct 13;24(10):1617-1626. doi: 10.1093/europace/euac081. PMID 35726877